CLINICAL TRIAL: NCT04919837
Title: The Efficacy of an Artificial Intelligence Platform to Adapt Visual Aids for Patients With Low Vision: a Randomised Controlled Trial
Acronym: AI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: 2nd Affilliated Hospital of Fujian Medical University (Unknown)
Responsible Party: Principal Investigator, Haotian Lin, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: SFLVRCT-2020
Record Dates: First submitted 2021-06-06; First posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-06

CONDITIONS: Ophthalmology; Low Vision Aids; Artificial Intelligence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Algorithm assisted group (Experimental): Patients receive assisting devices fitting services from human doctors assisted by the machine learning model
  Interventions: Other: Low vision aids
- Human doctor group (Experimental): Patients receive assisting devices fitting services from humanr doctors
  Interventions: Other: Low vision aids

INTERVENTIONS:
Other: Low vision aids — the assisting devices fitting for low-vision patients

SUMMARY:
According to the WHO's definition of visual impairment, as of 2018, there were approximately 1.3 billion people with visual impairment in the world, and only 10% of countries can provide assisting services for the rehabilitation of visual impairment. Although China is one of the countries that can provide rehabilitation services for patients with visual impairment, due to restrictions on the number of professionals in various regions, uneven diagnosis and treatment, and regional differences in economic conditions, not all visually impaired patients can get the rehabilitation of assisting device fitting.

Traditional statistical methods were not enough to solve the problem of intelligent fitting of assisting devices. At present, there are almost no intelligent fitting models of assisting devices in the world. Therefore, in order to allow more low-vision patients to receive accurate and rapid rehabilitation services, we conducted a cross-sectional study on the assisting devices fitting for low-vision patients in Fujian Province, China in the past five years, and at the same time constructed a machine learning model to intelligently predict the adaptation result of the basic assisting devices for low vision patients.

ELIGIBILITY:
Inclusion Criteria:

* Low vision Aged 3 to 105

Exclusion Criteria:

* Severe systemic diseases Failure to sign informed consent or unwilling to participate

Ages: 3 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-07-27 (Actual); Primary Completion 2021-07-27 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of giving up assisting devices | Baseline
  The investigator will calculate the proportion of giving up more than one assisting devices in two groups for three months and six months

SECONDARY OUTCOMES:
Time cost of using assisting devices of patients | Baseline
  The investigator will apply survival analysis for the time cost of using assisting devices in different groups.

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affilliated Hospital of Jujian Medical University, Quanzhou, Fujian, China